CLINICAL TRIAL: NCT06379659
Title: Effectiveness of Intrauterine Growth Hormone Infusion as an add-on Therapy to Conventional Hormone Therapy Compared to Placebo in Patients With Thin Endometrium Undergoing Frozen Thawed Embryo Transfer: A Double-blinded Parallel Exploratory Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Intrauterine Growth Hormone Administration as an add-on Therapy to Conventional Hormone Therapy Compared to Placebo in Patients With Thin Endometrium Undergoing Frozen Thawed Embryo Transfer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hatav Ghasemi Tehrani, Principal investigator, Associated professor of Infertility and In-Vivo-Fertilization, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.MUI.MED.REC.1402.449; IRCT20110908007513N18 (Registry Identifier: IRAN registry of clinical trials (IRCT))
Record Dates: First submitted 2024-04-11; First posted 2024-04-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Thin Endometrium; Infertility Female; Infertility
Keywords: Infertility; Infertility, Female; endometrial thickness; Thin Endoetrium; Growth Hormone; Human Growth Hormone; Somatropin; Intra-uterine infusion
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled exploratory clinical trial, controlled with a parallel placebo group and random allocation using an online based system.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In this study, a double-blind methodology will be employed to minimize bias. Patients will be administered medication without knowing the study group and placebo or treatment intervention. To ensure uniformity between growth hormone and placebo, which has a similar appearance to the placebo, will be prepared by an individual informed of the enrolled patients in the study and will be provided to the administering physician. The evaluator assessing outcomes such as clinical pregnancy rate and endometrial thickness will not know which treatment each patient received. Laboratory staff will also be unaware of the treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Growth hormone (Active Comparator)
  Interventions: Drug: Growh hormone
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Growh hormone — In this group, patients will receive growth hormone solution containing 1.99 milligrams of the drug dissolved in 1.5 milliliters of 0.9% saline solution (normal saline), in addition to standard hormonal therapy, starting from cycle day 10. Treatment sessions will be conducted at two-day intervals. In case of non-response to treatment (failure to reach a minimum endometrial thickness of 7 millimeters in the subsequent assessment), the patient will receive a maximum of 4 doses, and if response to treatment is observed, growth hormone infusion will be discontinued. All infusions will be administered intrauterinely via an Intrauterine Insemination (IUI) catheter.
  Arms: Growth hormone
Other: Placebo — Similar to the intervention group, from cycle day 10, an equal volume of 0.9% saline solution (normal saline) will be administered in addition to standard hormonal therapy. Treatment sessions will be conducted at two-day intervals. In case of non-response to treatment (failure to reach a minimum endometrial thickness of 7 millimeters in the subsequent assessment), the patient will receive a maximum of 4 doses, and if response to treatment is observed, placebo infusion will be discontinued. All infusions will be administered intrauterinely via an Intrauterine Insemination (IUI) catheter.
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to see if intrauterine growth hormone infusions can help subjects reach a suitable endometrial thickness in patients who are resistant to routine hormonal therapy for embryo transfer in the In Vitro Fertilization (IVF) cycle.

The primary aim of this study is to assess the effectiveness of injecting Growth hormone directly into the uterus to enhance endometrial thickness. Additionally, we aim to compare the likelihood of pregnancy between patients receiving the Growth hormone infusion and those receiving a placebo.

DETAILED DESCRIPTION:
Infertility impacts approximately 10-15% of couples globally, with over 1 million couples affected in Iran alone, adversely affecting their quality of life. However, Assisted Reproductive Technology (ART), notably In Vitro Fertilization (IVF), has markedly enhanced fertility outcomes for couples facing infertility.

The primary reason for IVF failure is often attributed to difficulties with embryo implantation. A crucial determinant in preparing the uterus for successful implantation is achieving an adequate endometrial thickness. A thin endometrium, typically defined as less than 7 mm in thickness, is associated with a significantly reduced likelihood of successful pregnancy following implantation. As a result, patients with thin endometrium are often deemed unsuitable candidates for implantation.

Despite exploring various pharmacological options, certain patients remain unable to achieve the minimum required endometrial thickness for successful implantation. Prior investigations have examined the impact of subcutaneous growth hormone injections on endometrial thickness in individuals with thin endometrium, yielding mixed results across studies. Direct infusion of drugs into the uterine cavity presents a potential route for localized treatment, thereby minimizing systemic effects under specific circumstances. Thus, different studies explored the possible intra-uterine effect of drugs such as Granulocyte colony stimulating factor (GCSF), and Human chorionic gonadotropin (hCG). To date, only an animal study and two small studies without control group have investigated the efficacy of direct intrauterine infusion of growth hormone in increasing endometrial thickness among patients with thin endometrium. However, the absence of randomized controlled trials with placebo groups limits our understanding of the effectiveness of intrauterine growth hormone therapy in this patient population. Thus, we aimed to design an exploratory randomized clinical trial with parallel placebo group to evaluate the effectiveness of intrauterine Growth Hormone infusion as an add-on therapy to conventional hormone therapy compared to placebo in patients with thin endometrium undergoing frozen thawed embryo transfer

ELIGIBILITY:
Inclusion Criteria:

* At least a history of cycle cancellation due to a thin endometrium less than 7 mm following standard hormonal treatment
* Availability of ≥1 embryo with good quality
* Normal baseline hormones value including: Testosterone, Progesterone, Prolactin, Luteinizing Hormone (LH), Follicle Stimulating Hormone (FSH)

Exclusion Criteria:

* Internal genital anomalies
* Active intrauterine infection Endometrial thickness≥7 on the 10th day of menstrual cycle
* History of Asherman syndrome
* History of cancer
* History of uterine surgery in past 3 months
* Intrauterine polyps visible in Transvaginal Ultrasonography
* Visible intrauterine adhesion
* Pathospermia in partner
* Premature ovarian failure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness | Baseline (On the 10th day of menstrual cycle), and On the day of response to treatment (in case of response) and in case of non-response to treatment on the 18th day of the mesntrual cycle
  Measurement of endometrial thickness will be performed utilizing transvaginal sonography due to its closer proximity to the endometrium and with an empty bladder. To minimize the potential bias of measuring endometrial thickness during uterus contraction, occur during contractions, measurements will be taken only after the patient's contractions have ceased.

SECONDARY OUTCOMES:
Clinical Pregnancy Rate | 6-8 of gestational week
  The number of fetuses that have a heartbeat and are not ectopic evaluated by Transvaginal Ultrasonography
Response to treatment | 2 days following the last dose of placebo or growth hormone
  The number of patients that reach at least 7 mm of endometrial thickness
Implantation rate | 6-8 of gestational week
  The number of gestational sacs to the number of transferred embryos evaluated by Transvaginal ultrasonography
IVF cancellation rate | 2 days following the last dose of placebo or growth hormone
  The number of patients who do not reach enough endometrial thickness for transferring despite maximum treatment
Early pregnancy complications | During the first 12 weeks of pregnancy
  Including early miscarriage (miscarriage in less than 12th gestational week) and Ectopic pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan Shahid Beheshti hospital, Hazrat e Maryam Fertility Center, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) may be shared following the publication of the study, as per specific requests from the researchers.

REFERENCES:
- [Result] Yu H, Gao S, Tang H, Chen H, Deng Z, Yang L, et al. Growth hormone intrauterine perfusion combined with replacement cycle in the treatment of non-response thin endometrium: report of 5 cases. Int J Clin Exp Med. 2016;9(6):11982-9
- [Result] Hosseini Aghdam S, Ghasemzadeh A, Farzadi L, Hamdi K, Baradaran-Binazir M, Nouri M, Fattahi A, Dttrich R. Growth Hormone: A Potential Treatment of Patients with Refractory Thin Endometrium: A Clinical Trial Study. Int J Fertil Steril. 2022 Oct 9;16(4):251-255. doi: 10.22074/ijfs.2022.541389.1210. PMID 36273309
- [Result] Li W, Cao Z, Yu X, Hu W. Effect of growth hormone on thin endometrium via intrauterine infusion. Ann Transl Med. 2021 Aug;9(16):1325. doi: 10.21037/atm-21-3583. PMID 34532462
- [Result] Altmae S, Aghajanova L. Growth Hormone and Endometrial Receptivity. Front Endocrinol (Lausanne). 2019 Sep 24;10:653. doi: 10.3389/fendo.2019.00653. eCollection 2019. PMID 31616379
- [Result] Liu KE, Hartman M, Hartman A. Management of thin endometrium in assisted reproduction: a clinical practice guideline from the Canadian Fertility and Andrology Society. Reprod Biomed Online. 2019 Jul;39(1):49-62. doi: 10.1016/j.rbmo.2019.02.013. Epub 2019 Mar 20. PMID 31029557
- [Result] Fu LL, Xu Y, Yan J, Zhang XY, Li DD, Zheng LW. Efficacy of granulocyte colony-stimulating factor for infertility undergoing IVF: a systematic review and meta-analysis. Reprod Biol Endocrinol. 2023 Apr 3;21(1):34. doi: 10.1186/s12958-023-01063-z. PMID 37013570